CLINICAL TRIAL: NCT06715553
Title: The Effect of Interventional Programs on Quality of Life and Functioning Among Patients With Schizophrenia
Brief Title: Interventional Programs' Impact on Patients' Quality of Life and Functioning
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Psychiatric Hospital of the Cross (Other)
Responsible Party: Principal Investigator, Marouan Zoghbi, Family medicine specialist, Hopital Psychiatrique De La Croix
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: HPC 001-08-2024
Record Dates: First submitted 2024-11-13; First posted 2024-12-04 (Actual); Last update posted 2025-03-10 (Actual); Status verified 2024-12

CONDITIONS: Schizophenia Disorder; Interventional Study
Keywords: schizophrenia; quality of life; Interventional program; Functional abilities
MeSH Terms: conditions — Schizophrenia | interventions — Reproductive Techniques, Assisted; Educational Status; Exercise; Nutritional Status

STUDY DESIGN:
Intervention Model Description: A 86 patients adhering to the inclusion and exclusion criteria will be randomized into two groups (43 patients in the intervention group and 43 patients in the control group) and the interventional model type will be in Parallel.
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Interventional group (Experimental): Participants will be randomly assigned to the intervention group
  Six types of intervention will be done on the patients as follows:
  * Psychoeducational intervention program prepared and will be applied by a psychologist
  * Art therapy program will be done by a psychologist
  * Bibliotherapy program will be done by a neuroscience person
  * Nutrition program will be done a nutritionist
  * Sport activity will be held by a physical trainee
  * Ping Pong activity will be done by a ping pong trainer
  Interventions: Behavioral: BALANCE Program (Body, Art, Learning, Activities, Nutrition, Creativity, and Education)
- Control Group (No Intervention): This group will follow the standard care provided by the hospital without any type of intervention

INTERVENTIONS:
Behavioral: BALANCE Program (Body, Art, Learning, Activities, Nutrition, Creativity, and Education) — Six types of intervention will be done on the patients as follows:
  * Psychoeducational intervention program
  * Art therapy program
  * Bibliotherapy program
  * Nutrition program
  * Sport activity
  * Ping Pong activity
  Arms: Interventional group

SUMMARY:
The objective of the study is to investigate the effect of interventional program in improving the quality of life for individuals with chronic schizophrenia The design of the study will be an interventional study - Randomized Control Trial - taking place in the Psychiatric hospital of the Cross Lebanon. Six types of intervention will be done on the patients such as ping-pong, sport exercise, psychoeducation program, nutrition, art therapy and bibliotherapy. A 100 patients adhering to the inclusion and exclusion criteria will be randomized into two groups (50 patients in the intervention group and 50 patients in the control group) - Simple Randomization. A Baseline and follow-up assessments will take place at the beginning of the study and after three months through using Arabic Validated Scales. The scales that be used are the following Positive and negative symptoms scale (PANSS), to determine severity of symptoms in patients. WHO quality of life questionnaire WHOQOL- BREF Arabic version: physical, psychological, social and environmental and EQ-5D scale, to determine quality of life of patients. MOCA scale to determine cognitive function, Rosenberg self-esteem questionnaire, Social functioning questionnaire QFS and Birchwood Insight Scale.

DETAILED DESCRIPTION:
Schizophrenia is considered to be one of the most disabling medical conditions in the world. It is characterized by a typical on-set in late adolescence to early adulthood, and a low remission rate, it is regarded as being a burden to patients' daily lives. Since there is evidence that the Quality of Life in patients with Schizophrenia is lower than the general population, it is believed that adhering to an interventional program might alleviate negative symptoms and cognitive deficits, leading to an improvement in Quality of Life.

Thus, this study will assess the impact of interventional program on improving the overall Quality of Life in patients with schizophrenia. Also, to assess the impact of the program on functional abilities, including occupational, social, and daily living skills, in patients with schizophrenia.

Participants will be recruited from the Psychiatric Hospital of the Cross. Eligible participants include individuals diagnosed with chronic schizophrenia, aged 18-65, and have given informed consent. To ensure the integrity and validity of the study, participants will be randomly assigned to either the intervention group or the control group (standard care) using randomized software.

By employing this randomization technique, we aim to minimize selection bias and ensure the comparability of the groups, thereby upholding the study's rigor and validity.

Intervention programs:

Six types of intervention will be done on the patients as follows:

* Psychoeducational intervention program prepared and will be applied by a psychologist
* Art therapy program will be done by a psychologist
* Bibliotherapy program will be done by a neuroscience person
* Nutrition program will be done a nutritionist
* Sport activity will be held by a physical trainee
* Ping Pong activity will be done by a ping pong trainer Data will be collected through direct observations, participant self-reports, and standardized assessments conducted by trained research staff.

ELIGIBILITY:
Inclusion Criteria:

* Individuals diagnosed with chronic schizophrenia according to DSM-V criteria
* Aged 18-65.
* Physically capable of participating in physical
* Clinically stable

Exclusion Criteria:

* Active substance use
* Severe cognitive impairment
* Intellectual disability

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 86 (Actual)
Dates: Start 2024-08-09 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
WHO Quality of Life-BREF (WHOQOL-BREF) | three months
  The WHOQOL-BREF measure the subjects' perception of QOL in every domain and the subjects' satisfaction with health and overall rating of QOL.
  The WHOQOL-BREF is a shortened version of the WHOQOL-100, it is composed of 26 items that uses a 5 point response scale ranging from 1 (very dissatisfied/very poor) to 5 (very satisfied/very good). Four domains were addressed including the physical health (seven items, Q3, Q4, Q10, Q15, Q16, Q17, Q18), psychological health (six items, Q5, Q6, Q7, Q11, Q19, Q26), social relations (three items, Q20, Q21, Q22), and environment (eight items, Q8, Q9, Q12, Q13, Q14, Q23, Q24, Q25).
  Domain scores are scaled in a positive direction (i.e. higher scores denote higher quality of life) with elevated score indicating higher quality of life. The mean score of items within each domain is used to calculate the domain score. Mean scores are then multiplied by 4 in order to make domain scores comparable with the scores used in the WHOQOL-100.
The 5-level EQ-5D version (EQ-5D-5L) | Three months
  The 5-level EQ-5D version (EQ-5D-5L) questionnaire is a globally used and multiply validated tool to assess health-related quality of life (HRQoL). It consists of 2 pages: the EQ-5D descriptive system and the EQ visual analogue scale (EQ VAS).
  The descriptive system comprises five dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Each dimension has 5 levels: no problems, slight problems, moderate problems, severe problems and extreme problems. The EQ VAS records the patient's self-rated health on a vertical visual analogue scale where the endpoints are labelled 'The best health you can imagine' and 'The worst health you can imagine'.

SECONDARY OUTCOMES:
Global Assessment of Functioning (GAF) | three months
  Global Assessment of Functioning (GAF) is a scoring system used to assess the severity of illness in psychiatry. It measures how much a person's symptoms affect their day-to-day life on a scale of 0 to 100. It is a numeric scale (0 through 100) used by mental health professionals and physicians to subjectively rate the social, occupational, and psychological functioning of adults. The highest ratings are 91-100, "Superior functioning in a wide range of activities and the lowest ratings (besides a 0, for "Inadequate information") are 1-10, "Persistent danger of severely hurting self or others…OR persistent inability to maintain minimal personal hygiene OR serious suicidal act with clear expectation of death.
Questionnaire du focntionnement sociale (QFS) | three months
  Questionnaire du focntionnement sociale (QFS) It is a brief self-assessment questionnaire made up of 16 questions covering the general functioning in the last 15 days. Eight questions assess the frequency of social behaviors, and the eight other questions focus on satisfaction that is withdrawn from these behaviors. The QFS makes it possible to calculate three main indices: a "Frequency" index, a "Satisfaction" index and a "Global" index, which corresponds to the sum of the two previous ones. The "Frequency" and "Satisfaction" index scores range from 8 to 40 while the "Overall" index score ranges from 16 to 80. A higher score corresponds to a better level of functioning.

OTHER OUTCOMES:
Clinical symptoms | three months
  Positive and Negative Syndrome Scale (PANSS) The PANSS is a scale validated in Lebanon that evaluate the clinical symptoms of the patients. It consists of 30 items, divided into 3 subcomponents: positive symptoms (seven items: P1-P7), negative symptoms (seven items: N1- N7) and symptoms of general psychopathology (16 items: G1-G16). All items are scored with values from 1 to 7, with 1 reflecting no symptoms and 7 reflecting extremely severe symptoms. The scores of these scales are calculated by the sum of the elements of each component [15]. The score for the positive and negative scales varies between 7 and 49 while the score varies from 16 to 112 for the general psychopathology scale. The total score is obtained by the sum of all the items

CONTACTS AND LOCATIONS:
Locations (1):
- Psychiatric Hospital of the Cross, Beirut, Lebanon

IPD SHARING:
Plan to Share IPD: Undecided
The psychiatric patients is considered as a vulnerable population and at this time we respectfully request no to share personal data although anonymous.

REFERENCES:
- [Background] Deenik J, Tenback DE, van Driel HF, Tak ECPM, Hendriksen IJM, van Harten PN. Less Medication Use in Inpatients With Severe Mental Illness Receiving a Multidisciplinary Lifestyle Enhancing Treatment. The MULTI Study III. Front Psychiatry. 2018 Dec 18;9:707. doi: 10.3389/fpsyt.2018.00707. eCollection 2018. PMID 30618878
- [Background] Effect of psycho-educational intervention on drug adherence and quality of life among patients with Schizophrenia in Jigawa State, Nigeria
- [Background] Hjorth P, Medici CR, Juel A, Madsen NJ, Vandborg K, Munk-Jorgensen P. Improving quality of life and physical health in patients with schizophrenia: A 30-month program carried out in a real-life setting. Int J Soc Psychiatry. 2017 Jun;63(4):287-296. doi: 10.1177/0020764017702172. Epub 2017 Apr 3. PMID 28367717
- [Background] Kang R, Wu Y, Li Z, Jiang J, Gao Q, Yu Y, Gao K, Yan Y, He Y. Effect of Community-Based Social Skills Training and Tai-Chi Exercise on Outcomes in Patients with Chronic Schizophrenia: A Randomized, One-Year Study. Psychopathology. 2016;49(5):345-355. doi: 10.1159/000448195. Epub 2016 Sep 2. PMID 27584836
- See also: The link describe the study site where the protocol is being applied. — http://www.hopitalpsychiatriquedelacroix.org.lb/french/